CLINICAL TRIAL: NCT03761667
Title: Usefulness of Narrow Band Imaging (NBI) for Complete Endoscopic Resection of Sessile Serrated Adenoma/Polyp (SSA/P): NASA Study
Brief Title: Usefulness of NBI for Complete Endoscopic Resection of SSA/P
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Soonchunhyang University Hospital (Other)
Responsible Party: Principal Investigator, Hyun Gun, Kim. M.D., Ph.D., Associate professor, Soonchunhyang University Hospital
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: NASA
Record Dates: First submitted 2018-11-29; First posted 2018-12-03 (Actual); Last update posted 2018-12-03 (Actual); Status verified 2018-11

CONDITIONS: Sessile Serrated Adenoma/Polyps
MeSH Terms: conditions — Polyps

ARMS (2):
- NBI (Experimental): The group of NBI inspection on resection margin for surveillance of remnant tissue of SSA/P right after the endoscopic resection. If the remnant tissue is detected using NIB inspection, additional endoscopic resection should be performed.
  Interventions: Other: Endoscopy using Narrow band imaging
- White light endoscopy (WLE) (No Intervention): The group of WLE inspection on resection margin for surveillance of remnant tissue of SSA/P right after the endoscopic resection. If the remnant tissue is detected using NIB inspection, additional endoscopic resection should be performed.

INTERVENTIONS:
Other: Endoscopy using Narrow band imaging — Inspection of resection margin of SSA/P for the evaluation of complete resection or the presence of remnant lesion using NBI method
  Arms: NBI

SUMMARY:
This study is a prospective randomized study to evaluate the role of NBI for improving complete resection rate of sessile serrated adenoma/polyp (SSA/P). The authors will enroll consecutive patients who underwent colon polypectomy for SSA/P during colonoscopy. The authors will inspect resection margin of SSA/P using white light endosocpy (WLE) or NBI after randomization for the evaluation of remnant lesion. Additional resection will be performed for suspicious of remnant lesion, and then 4 biopsies from 4 quadrants of margin for evaluation of complete resection.

DETAILED DESCRIPTION:
This study is a prospective randomized multi-center study to evaluate the role of NBI for improving complete resection rate of sessile serrated adenoma/polyp (SSA/P).

The authors will enroll consecutive patients who underwent colon polypectomy for suspicious SSA/P during colonoscopy.

All patients who undergo polypectomy will be enrolled, but excluded as follows; 1. poor bowel preparation according to Boston bowel preparation scale calculation, 2. inflammatory bowel disease, 3. failure of cecal insertion, 4. continuous anti-plate agents or anti-coagulation agents users.

First, the authors will inspect polyp using the arbitrary endoscopic criteria by inspection of white light endoscopy (WLE) and if that lesion is satisfied with 3 or more than 3 out of 5 categories (1. located in the right colon, 2. flat shape, 3. covered with mucus cap or debris, 4. 1 cm or larger than 1 cm in size, 5. varicose superficial vessel was seen on the surface after submucosal injection), endoscopic resection will be performed.

And then, the authors will inspect the resection margin carefully using NBI or WLE by pre-randomization before endoscopic resection. If the remnant tissue is detected, additional endoscopic resection will be performed.

ed margin as two groups (NBI inspection group and WLE inspection

And then, 4 biopsies from 4 quadrants of margin for evaluation of complete resection.

Primary end-point is comparing the rate of additional resection for remnant lesion, the SSA/P diagnosis rate of the remnant lesions after the additional resection, and the complete resection rate of the target lesion between two groups.

Secondary aim is evaluate the accuracy for SSA/P using arbitrary WLE criteria. For evaluation of the accuracy of arbitrary WLE criteria, the authors will compare the pathologic diagosis rate of SSA/P for each criterion, and calculate the sensitivity, the specificity, the positive predictive value, the negative predictive value, and the accuracy with area under curve of ROC.

The authors hypothesized complete resection rate of SSA/P as 90% in the NBI inspection group and 70% in the WLE inspection group based on previous studies including CARE study.

The sample size was calculated as 118 (each 59) patients of SSA/P. Study duration will be 2 years.

ELIGIBILITY:
Inclusion Criteria:

* Colonoscopy examinee with suspicious SSA/P

Exclusion Criteria:

* Poor bowel preparation (total Boston bowel preparation scale < 6 or any region score < 2)
* Inflammatory bowel disease
* failed cecal insertion of colonoscopy
* continuous taking anticoagulation or anti-platelet drugs until on the procedure day

Sex: All | Healthy Volunteers: Yes
Age Groups: Child, Adult, Older Adult
Enrollment: 118 (Actual)
Dates: Start 2015-12-23 (Actual); Primary Completion 2018-11-10 (Actual); Study Completion 2018-11-25 (Actual)

PRIMARY OUTCOMES:
the detection rate of remnant lesion, | 2 years after IRB
  Comparing the detection rate of remnant SSA/P right after the endoscopic resection
The diagnosis rate of SSA/P in the remnant tissue | 2 years after IRB
  Pathologic diagnosis rate of SSA/P after the additional endoscopic resection of the remnant tissue detected by NBI or WLE right after the endoscopic resection.
Incomplete resection rate of SSA/P | 2 years after IRB
  Compare the incomplete resection rate of SSA/P using four directional biopsied on the resection margin after the endoscopic resection including additional resection

SECONDARY OUTCOMES:
Accuracy of arbitrary endoscopic criteria for SSA/P inspection by white light endoscopy | 2 years after IRB
  In this study, the authors made the arbitrary endoscopic criteria for suspicion of SSA/P by inspection of WLE.